CLINICAL TRIAL: NCT02916485
Title: BIOTRONIK - Safety and Clinical Performance Of the Magmaris Drug Eluting Absorbable Metal Scaffold in a Cohort of Patients in India With de Novo Lesions in NatiVE Coronary Arteries
Brief Title: Safety and Clinical Performance of a Sirolimus-eluting Absorbable Metal Scaffold
Acronym: BIOSOLVE-India
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting National Pharmaceutical Pricing Authority (NPPA) review of ceiling prices for innovative products in India.
Sponsor: Biotronik AG (Industry)
Collaborators: CBCC-VIBGYOR Research Pvt. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1601
Record Dates: First submitted 2016-09-23; First posted 2016-09-27 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Coronary Artery Disease
Keywords: bioresorbable scaffold; vascular restoration therapy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bioresorbable scaffold (Experimental): Percutaneous coronary intervention (PCI) with a sirolimus-eluting resorbable coronary magnesium scaffold
  Interventions: Device: Bioresorbable scaffold

INTERVENTIONS:
Device: Bioresorbable scaffold — Percutaneous coronary intervention (PCI)
  Other Names: Sirolimus-eluting resorbable coronary magnesium scaffold; Magmaris

SUMMARY:
Assessment of the clinical performance and the safety of the Magmaris Sirolimus-Eluting Resorbable Coronary Magnesium Scaffold in a cohort of patients in India with de novo coronary artery lesions.

DETAILED DESCRIPTION:
This is a prospective, multi-centre, single-arm, open label trial to assess the safety and clinical performance of Magmaris Drug Eluting Absorbable Metal Scaffold.

A total of up to 110 patients with de novo lesions in native coronary arteries will be enrolled at up to 8 investigational sites in India.

In-hospital clinical follow-up visits will take place at 1 and 6 months post procedure.

The primary endpoint is target lesion failure (a composite of cardiac death, target vessel Q-wave or non-Q wave myocardial infarction, coronary artery bypass grafting, clinically driven target lesion revascularization) at 1 month post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years and ≤ 80 years of age
2. Written subject informed consent available prior to percutaneous coronary intervention (PCI). Remark: Vulnerable subjects may not be enrolled in this trial
3. Subject with stable or unstable angina pectoris or documented silent ischemia
4. Subject eligible for PCI
5. Subject acceptable candidate for coronary artery bypass surgery
6. Subject with a maximum of two single de novo lesions in two different major epicardial vessels
7. Reference vessel diameter between 2.7-3.7 mm by visual estimation, depending on the scaffold size used
8. Target lesion length ≤ 21 mm by visual estimation, depending on the scaffold size used
9. Target lesion stenosis by visual estimation ≥ 50% - < 100% and TIMI flow ≥1
10. Eligible for Dual Anti Platelet Therapy (DAPT)

Exclusion Criteria:

1. Pregnant or breast-feeding females or females who intend to become pregnant during the time of the study
2. Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation myocardial infarction (STEMI) within 72 hours prior to the index procedure. Note: Hemodynamically stable non-STEMI (NSTEMI) subjects are eligible for study enrollment
3. Subjects with a ≥2 fold CK level or in absence of CK a ≥3 fold CKMB level above the upper range limit within 24 hours prior to the index procedure
4. Left main coronary artery disease
5. Three-vessel coronary artery disease at time of procedure
6. Thrombus in target vessel
7. Subject is currently participating in another study with an investigational device or an investigational drug and has not reached the primary endpoint yet
8. Planned interventional treatment of any non-target vessel within 30 days post-procedure
9. Subject is on dialysis
10. Planned intervention of the target vessel after the index procedure
11. Ostial target lesion (within 3.0 mm of vessel origin)
12. Target lesion involves a side branch >2.0 mm in diameter
13. Documented left ventricular ejection fraction (LVEF) ≤ 30%
14. Heavily calcified lesion
15. Target lesion is located in or supplied by an arterial or venous bypass graft
16. The target lesion requires treatment with a device other than the pre-dilatation balloon prior to the Magmaris study device placement (including but not limited to directional coronary atherectomy, excimer laser, rotational atherectomy, etc.)
17. Unsuccessful pre-dilatation, defined as minimal lumen diameter smaller than the respective crossing profile of the Magmaris study device and angiographic complications (e.g. distal embolization, side branch closure, extensive dissections that can't be covered by a single scaffold), by visual estimation
18. Known allergies to: Acetylsalicylic Acid (ASA), Heparin, contrast medium, Sirolimus, Everolimus or similar drugs (i.e., ABT 578, Biolimus, Tacrolimus), PLLA, Silicon Carbide, Magnesium, Yttrium, Neodymium, Zirconium, Gadolinium, Dysprosium, Tantalum
19. Impaired renal function (serum creatinine > 2.5 mg/dl or 221 µmol/l) determined within 72 hours prior to index procedure
20. Subject is receiving oral or intravenous immunosuppressive therapy (inhaled steroids are not excluded) or has known life limiting immunosuppressive or autoimmune disease (e.g.,human immunodeficiency virus, systemic lupus erythematosus, but not including diabetes mellitus)
21. Proximal or distal to the target lesion located stenosis that might require future revascularization or impede run off detected during diagnostic angiography
22. Life expectancy less than 6 months
23. Planned surgery or dental surgical procedure within 6 months after index procedure
24. Subject with tortuous vessel that may impair scaffold placement in the region of obstruction or proximal to the lesion
25. In the investigators opinion subjects will not be able to comply with the follow-up requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 1 month post-procedure
  TLF is a composite of cardiac death, target vessel Q-wave or non-Q wave myocardial infarction (MI), coronary artery bypass graft (CABG), clinically driven target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Target lesion failure (TLF) | 6 months post-procedure
  TLF is a composite of cardiac death, target vessel Q-wave or non-Q wave myocardial infarction (MI), coronary artery bypass graft (CABG), clinically driven target lesion revascularization (TLR)
Target vessel failure (TVF) | 1 and 6 months post-procedure
  TVF is a composite of cardiac death, target vessel Q-wave or non-Q wave myocardial infarction (MI), coronary artery bypass graft (CABG), clinically driven target vessel revascularization (TVR)
Clinically driven target lesion revascularization | 1 and 6 months post-procedure
Cardiac death | 1 and 6 months post-procedure
Myocardial infarction | 1 and 6 months post-procedure
Scaffold thrombosis | 1 and 6 months post-procedure
  Scaffold thrombosis is composite of definite and probable scaffold thrombosis according to ARC definition
Incidence of procedure success | 3 days (plus or minus 2 days)
  Procedure Success is a composite of achievement of a final diameter stenosis of <30% by visual assessment or on-line quantitative coronary angiography, without the occurrence of death, Q-wave or non-Q-wave MI, or repeat revascularization of the target lesion during the hospital stay (3 days plus or minus 2 days)
Incidence of device success | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
  Device Success is a composite of a final residual diameter stenosis of <30% by visual assessment or on-line quantitative coronary angiography, using the assigned device only, successful delivery of the scaffold to the target lesion site in the coronary artery, appropriate scaffold deployment, successful removal of the device, safe removal of the device in case of deployment failure.

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences, Delhi, India

IPD SHARING:
Plan to Share IPD: No